CLINICAL TRIAL: NCT00996658
Title: A Phase III, Randomised, Double Blind, Placebo Controlled Parallel Group Efficacy and Safety Study of Linagliptin 5 mg Administered Orally Once Daily Over 24 Weeks in Type 2 Diabetic Patients With Insufficient Glycaemic Control Despite a Therapy of Metformin in Combination With Pioglitazone
Brief Title: Linagliptin Versus Placebo in Type 2 Diabetic Patients With Inadequate Glycaemic Control on Metformin in Combination With Pioglitazone
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1218.61; 2009-013289-20 (EudraCT Number: EudraCT)
Record Dates: First submitted 2009-10-15; First posted 2009-10-16 (Estimated); Results first posted 2013-03-26 (Estimated); Last update posted 2014-03-26 (Estimated); Status verified 2014-02

CONDITIONS: Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Linagliptin

ARMS (2):
- Linagliptin (Experimental): Linagliptin tablets once daily
  Interventions: Drug: Linagliptin
- Placebo (Placebo Comparator): Placebo tablets once daily
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Placebo — Placebo matching linagliptin tablets once daily
  Arms: Placebo
Drug: Linagliptin — Linagliptin tablets once daily
  Arms: Linagliptin

SUMMARY:
The objective of the current study is to investigate the efficacy, safety and tolerability of Linagliptin (5 mg once daily) compared to placebo given for 24 weeks as add on therapy to metformin in combination with pioglitazone in patients with type 2 diabetes mellitus with insufficient glycaemic control.

ELIGIBILITY:
Inclusion criteria:

1. Diagnosis of diabetes mellitus prior to informed consent
2. Patients treated with metformin and pioglitazone (therapy should be unchanged for 12 weeks)
3. Glycosylated haemoglobin A1 >= 7.5% and <= 10%
4. Age between 18 and less than 80
5. - Body Mass index less or equal to 45

Exclusion criteria:

1. Uncontrolled hyperglycaemia during run in period
2. Myocardial infarction, stroke or transient ischaemic accident within 3 months prior to informed consent
3. Impaired hepatic function
4. Gastric by pass surgery
5. Treatment with roziglitazone, GLP 1 analogues, DPP-4 inhibitors or insulin within 3 months prior to informed consent
6. Treatment with anti-obesity drugs
7. Current treatment with systemic steroids at the time of informed consent or change in dosage of thyroid hormones within 6 weeks prior to informed consent
8. Premenopausal women who are nursing or pregnant or are of child-bearing potential and are not practicing an acceptable method of birth control or do not plan to continue using this method during the trial

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 278 (Actual)
Dates: Start 2009-10; Primary Completion 2012-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (52):
- United States (29):
  - 1218.61.01028 Boehringer Ingelheim Investigational Site, Escondido, California
  - 1218.61.01014 Boehringer Ingelheim Investigational Site, Greenbrae, California
  - 1218.61.01015 Boehringer Ingelheim Investigational Site, Los Angeles, California
  - 1218.61.01042 Boehringer Ingelheim Investigational Site, Paramount, California
  - 1218.61.01046 Boehringer Ingelheim Investigational Site, Poway, California
  - 1218.61.01044 Boehringer Ingelheim Investigational Site, San Diego, California
  - 1218.61.01009 Boehringer Ingelheim Investigational Site, Miami, Florida
  - 1218.61.01049 Boehringer Ingelheim Investigational Site, Lawrenceville, Georgia
  - 1218.61.01008 Boehringer Ingelheim Investigational Site, Roswell, Georgia
  - 1218.61.01040 Boehringer Ingelheim Investigational Site, Meridian, Idaho
  - 1218.61.01016 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1218.61.01018 Boehringer Ingelheim Investigational Site, Chicago, Illinois
  - 1218.61.01048 Boehringer Ingelheim Investigational Site, Lafayette, Indiana
  - 1218.61.01001 Boehringer Ingelheim Investigational Site, Auburn, Maine
  - 1218.61.01043 Boehringer Ingelheim Investigational Site, Olive Branch, Mississippi
  - 1218.61.01052 Boehringer Ingelheim Investigational Site, Las Vegas, Nevada
  - 1218.61.01030 Boehringer Ingelheim Investigational Site, New York, New York
  - 1218.61.01007 Boehringer Ingelheim Investigational Site, Greensboro, North Carolina
  - 1218.61.01004 Boehringer Ingelheim Investigational Site, Jacksonville, North Carolina
  - 1218.61.01023 Boehringer Ingelheim Investigational Site, Wilmington, North Carolina
  - 1218.61.01027 Boehringer Ingelheim Investigational Site, Perrysburg, Ohio
  - 1218.61.01031 Boehringer Ingelheim Investigational Site, East Providence, Rhode Island
  - 1218.61.01017 Boehringer Ingelheim Investigational Site, Simpsonville, South Carolina
  - 1218.61.01005 Boehringer Ingelheim Investigational Site, Dallas, Texas
  - 1218.61.01006 Boehringer Ingelheim Investigational Site, Houston, Texas
  - 1218.61.01053 Boehringer Ingelheim Investigational Site, San Antonio, Texas
  - 1218.61.01003 Boehringer Ingelheim Investigational Site, Sugar Land, Texas
  - 1218.61.01024 Boehringer Ingelheim Investigational Site, Bennington, Vermont
  - 1218.61.01020 Boehringer Ingelheim Investigational Site, Spokane, Washington
- France (9):
  - 1218.61.3301A Boehringer Ingelheim Investigational Site, Besançon
  - 1218.61.3306A Boehringer Ingelheim Investigational Site, Béziers
  - 1218.61.3311A Boehringer Ingelheim Investigational Site, Béziers
  - 1218.61.3309A Boehringer Ingelheim Investigational Site, Bourg Des Cptes
  - 1218.61.3310A Boehringer Ingelheim Investigational Site, Cournonterral
  - 1218.61.3312A Boehringer Ingelheim Investigational Site, Laval
  - 1218.61.3313A Boehringer Ingelheim Investigational Site, Louvigné-de-Bais
  - 1218.61.3305A Boehringer Ingelheim Investigational Site, Paris
  - 1218.61.3307A Boehringer Ingelheim Investigational Site, Paris
- India (11):
  - 1218.61.91002 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.61.91003 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.61.91004 Boehringer Ingelheim Investigational Site, Bangalore
  - 1218.61.91008 Boehringer Ingelheim Investigational Site, Hyderabad
  - 1218.61.91009 Boehringer Ingelheim Investigational Site, Jaipur
  - 1218.61.91010 Boehringer Ingelheim Investigational Site, Karnataka
  - 1218.61.91001 Boehringer Ingelheim Investigational Site, Maharashtra
  - 1218.61.91006 Boehringer Ingelheim Investigational Site, Maharashtra
  - 1218.61.91011 Boehringer Ingelheim Investigational Site, Maharashtra
  - 1218.61.91005 Boehringer Ingelheim Investigational Site, Mumbai
  - 1218.61.91007 Boehringer Ingelheim Investigational Site, Mumbai
- Philippines (3):
  - 1218.61.63003 Boehringer Ingelheim Investigational Site, Cebu City
  - 1218.61.63004 Boehringer Ingelheim Investigational Site, Cebu City
  - 1218.61.63002 Boehringer Ingelheim Investigational Site, Davao City

REFERENCES:
- [Derived] Bajaj M, Gilman R, Patel S, Kempthorne-Rawson J, Lewis-D'Agostino D, Woerle HJ. Linagliptin improved glycaemic control without weight gain or hypoglycaemia in patients with type 2 diabetes inadequately controlled by a combination of metformin and pioglitazone: a 24-week randomized, double-blind study. Diabet Med. 2014 Dec;31(12):1505-14. doi: 10.1111/dme.12495. Epub 2014 Jul 7. PMID 24824197

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo Tablet: Placebo matching linagliptin 5 mg tablet
- Linagliptin 5 mg Tablet: Linagliptin 5 mg (milligrams) tablet given by mouth once daily
Period: Overall Study
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Started | 92 | 186
Completed | 76 | 165
Not Completed | 16 | 21
Not completed — Adverse Event | 2 | 5
Not completed — Protocol Violation | 0 | 1
Not completed — Lost to Follow-up | 2 | 5
Not completed — Non-compliance issues | 3 | 3
Not completed — Other | 9 | 7

BASELINE CHARACTERISTICS:
Population: Six participants (three participants per treatment) were excluded from all analyses due to serious site non-compliance. Thus, the total participants in Baseline Measures (272) is six less than total in Participant Flow (278).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet | Total
Number analyzed (Participants) | 89 | 183 | 272
Age, Continuous [Mean (Standard Deviation); unit: years] | 55.2 (8.4) | 53.1 (9.7) | 53.8 (9.3)
Age, Customized [Number; unit: participants]
  < 65 years | 79 | 162 | 241
  65 to 74 years | 8 | 20 | 28
  >= 75 years | 2 | 1 | 3
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 40 | 100 | 140
  Male | 49 | 83 | 132
Weight [Mean (Standard Deviation); unit: kilograms] | 74.4 (19.8) | 74.4 (20.4) | 74.4 (20.2)
Weight categories [Number; unit: participants]
  <= 70 kilograms | 46 | 97 | 143
  > 70 to 80 kilograms | 17 | 32 | 49
  > 80 to 90 kilograms | 10 | 18 | 28
  > 90 kilograms | 16 | 36 | 52
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilograms per square meter] | 28.1 (5.5) | 28.2 (5.2) | 28.2 (5.3)
Body Mass Index (BMI) categories [Number; unit: participants]
  < 25 kilograms/square meter | 29 | 51 | 80
  >= 25 and < 30 kilograms/square meter | 38 | 76 | 114
  >= 30 kilograms/square meter | 22 | 56 | 78
Height [Mean (Standard Deviation); unit: centimeters] | 162.0 (11.0) | 161.4 (11.4) | 161.6 (11.2)
Waist circumference [Mean (Standard Deviation); unit: centimeters] | 97.7 (13.5) | 98.1 (13.1) | 98.0 (13.2)
Smoking status [Number; unit: participants]
  Never smoked | 75 | 151 | 226
  Ex-smoker | 12 | 16 | 28
  Currently smokes | 2 | 16 | 18
Alcohol status [Number; unit: participants]
  Non drinker | 79 | 156 | 235
  Drinks - no interference with study | 10 | 27 | 37
  Drinks - investigator opinion/interfere with study | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in HbA1c (Glycosylated Hemoglobin) After 24 Weeks
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin
Time Frame: baseline, 24 weeks
Population: Full Analysis Set (FAS) includes all randomized patients who received study medication and had both a baseline HbA1c value and an on-treatment HbA1c value. Three subjects in each arm excluded for site non-compliance.
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 89 | 179
Percentage | -0.27 (0.13) | -0.84 (0.11)
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model included terms for treatment, baseline HbA1c and centre; Mean Difference (Final Values) = -0.57, 95% CI [-0.83 to -0.31]

2. Secondary Outcome: Change From Baseline in HbA1c (Glycosylated Hemoglobin) After 6 Weeks
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin
Time Frame: baseline, 6 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 89 | 179
Percentage | -0.19 (0.11) | -0.60 (0.09)
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model included terms for treatment, baseline HbA1c and centre; Mean Difference (Final Values) = -0.41, 95% CI [-0.61 to -0.21]

3. Secondary Outcome: Change From Baseline in HbA1c (Glycosylated Hemoglobin) After 12 Weeks
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin
Time Frame: baseline, 12 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 89 | 179
Percentage | -0.28 (0.12) | -0.82 (0.10)
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model included terms for treatment, baseline HbA1c and centre; Mean Difference (Final Values) = -0.54, 95% CI [-0.79 to -0.28]

4. Secondary Outcome: Change From Baseline in HbA1c (Glycosylated Hemoglobin) After 18 Weeks
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin
Time Frame: baseline, 18 weeks
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Percentage
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 89 | 179
Percentage | -0.37 (0.12) | -0.91 (0.10)
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p < 0.0001, ANCOVA; ANCOVA model included terms for treatment, baseline HbA1c and centre; Mean Difference (Final Values) = -0.54, 95% CI [-0.80 to -0.29]

5. Secondary Outcome: Occurrence of Absolute Efficacy Response (HbA1c < 7%) After 24 Weeks
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin
Time Frame: 24 weeks
Population: Full Analysis Set (FAS) includes all randomized patients who received study medication and had HbA1c >=7.0% at baseline (NCF). Three subjects in each arm excluded for site non-compliance.
Measure: Number; unit: Participants
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 87 | 176
Participants
  Responder (HbA1c < 7.0%) | 12 | 57
  Non-responder (HbA1c >= 7.0%) | 75 | 118
  Missing | 0 | 1
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Linagliptin vs Placebo; Test type: Superiority or Other; p = 0.0033, Regression, Logistic; Odds Ratio (OR) = 2.939, 95% CI 2-sided [1.432 to 6.032]

6. Secondary Outcome: Occurrence of Absolute Efficacy Response (HbA1c < 6.5%) After 24 Weeks
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin
Time Frame: 24 weeks
Population: Full Analysis Set (FAS) includes all randomized patients who received study medication and had HbA1c >=6.5% at baseline (NCF). Three subjects in each arm excluded for site non-compliance.
Measure: Number; unit: Participants
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 89 | 178
Participants
  Responder (HbA1c < 6.5%) | 5 | 34
  Non-responder (HbA1c >= 6.5%) | 84 | 143
  Missing | 0 | 1
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Linagliptin vs Placebo; Test type: Superiority or Other; p = 0.0074, Regression, Logistic; Odds Ratio (OR) = 3.902, 95% CI 2-sided [1.440 to 10.572]

7. Secondary Outcome: Occurrence of Relative Efficacy Response (Reduction in HbA1c >= 0.5%) After 24 Weeks
Description: Glycosylated hemoglobin is reported as a percentage of the total hemoglobin
Time Frame: 24 weeks
Population: Full Analysis Set (FAS) includes all randomized patients who received study medication. Three subjects in each arm excluded for site non-compliance.
Measure: Number; unit: Participants
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 89 | 179
Participants
  Responder (reduction in HbA1c >= 0.5%) | 44 | 117
  Non-responder (reduction in HbA1c < 0.5%) | 45 | 61
  Missing | 0 | 1
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Linagliptin vs. Placebo; Test type: Superiority or Other; p = 0.0071, Regression, Logistic; Odds Ratio (OR) = 2.059, 95% CI 2-sided [1.216 to 3.485]

8. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) After 24 Weeks
Description: Adjusted mean change in fasting plasma glucose (FPG) from baseline at week 24
Time Frame: baseline, 24 weeks
Population: Full Analysis Set (FAS) includes all randomized patients who received study medication and had both a baseline FPG value and an on-treatment FPG value. Three subjects in each arm excluded for site non-compliance.
Measure: Least Squares Mean (Standard Error); unit: mg/dL (milligrams per deciliter)
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 86 | 175
mg/dL (milligrams per deciliter) | 0.1 (3.8) | -10.3 (2.7)
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p = 0.0280, ANCOVA; ANCOVA model included terms for treatment, baseline HbA1c, baseline FPG, and centre; Mean Difference (Final Values) = -10.4, 95% CI [-19.6 to -1.1]

9. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) After 6 Weeks
Description: Adjusted mean change in fasting plasma glucose (FPG) from baseline at week 6
Time Frame: baseline, 6 weeks
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: mg/dL (milligrams per deciliter)
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 86 | 175
mg/dL (milligrams per deciliter) | 12.4 (5.4) | -3.3 (4.6)
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p = 0.0006, ANCOVA; ANCOVA model included terms for treatment, baseline HbA1c, baseline FPG, and centre; Mean Difference (Final Values) = -15.7, 95% CI [-24.5 to -6.8]

10. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) After 12 Weeks
Description: Adjusted mean change in fasting plasma glucose (FPG) from baseline at week 12
Time Frame: baseline, 12 weeks
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: mg/dL (milligrams per deciliter)
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 86 | 175
mg/dL (milligrams per deciliter) | 3.8 (4.6) | -7.1 (3.6)
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p = 0.0210, ANCOVA; ANCOVA model included terms for treatment, baseline HbA1c, baseline FPG, and centre; Mean Difference (Final Values) = -10.9, 95% CI [-20.2 to -1.7]

11. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) After 18 Weeks
Description: Adjusted mean change in fasting plasma glucose (FPG) from baseline at week 18
Time Frame: baseline, 18 weeks
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: mg/dL (milligrams per deciliter)
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Number analyzed (Participants) | 86 | 175
mg/dL (milligrams per deciliter) | -2.4 (4.1) | -8.6 (2.8)
Statistical Analysis 1: Comparison: Placebo Tablet vs Linagliptin 5 mg Tablet; Test type: Superiority or Other; p = 0.2137, ANCOVA; ANCOVA model included terms for treatment, baseline HbA1c, baseline FPG, and centre; Mean Difference (Final Values) = -6.2, 95% CI [-16.0 to 3.6]

ADVERSE EVENTS:
Time Frame: From drug start up to drug stop (max 24 weeks)+ 7 days
Description: For the analysis of AEs, all events with an onset after the first dose of trial medication up to a period of 7 days after the last dose of trial medication were assigned to the randomised treatment period.
Arm/Group | Placebo Tablet | Linagliptin 5 mg Tablet
Serious Adverse Events (participants affected / at risk) | 3/89 | 4/183
Other Adverse Events (participants affected / at risk) | 16/89 | 31/183
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Tablet (N=89) | Linagliptin 5 mg Tablet (N=183)
Anaemia (Blood and lymphatic system disorders) | 0 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Cataract (Eye disorders) | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1
Hepatitis E (Infections and infestations) | 1 | 0
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Calculus bladder (Renal and urinary disorders) | 0 | 1
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo Tablet (N=89) | Linagliptin 5 mg Tablet (N=183)
Anaemia (Blood and lymphatic system disorders) | 6 | 13
Hyperglycaemia (Metabolism and nutrition disorders) | 7 | 11
Hypoglycaemia (Metabolism and nutrition disorders) | 4 | 10

LIMITATIONS AND CAVEATS:
During the conduct of this trial, pioglitazone was removed from the market in France due to safety issues, and this resulted in premature termination of a number of French patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.